CLINICAL TRIAL: NCT05054452
Title: Predicting Fluid Responsiveness in Mechanically Ventilated Critically Ill Children and Neonates Using Transthoracic Echocardiography
Brief Title: Predicting Fluid Responsiveness in Mechanically Ventilated Critically Ill Children Using Transthoracic Echocardiography
Acronym: PREDIPEN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-A00203-38
Record Dates: First submitted 2021-06-21; First posted 2021-09-23 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-09

CONDITIONS: Fluid Therapy; Hemodynamics; Hypovolemia; Shock
Keywords: children; critically ill; fluid therapy; fluid responsiveness; hemodynamics; hypovolemia; shock; echocardiography
MeSH Terms: conditions — Hypovolemia; Shock; Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Echocardiographic assessment (Experimental): At baseline before standardized volume expansion, a first set of echocardiographic measurements will be performed. Then, we will perform 15-second end-expiratory and end-inspiratory occlusions. Occlusions will be separated by 1 minute to allow the cardiac index to return to its baseline value. A last set of measurements will be performed after fluid administration. Ventilatory settings and other treatments will remain unchanged during the study period.
  Interventions: Device: Echocardiographic assessment

INTERVENTIONS:
Device: Echocardiographic assessment — At baseline before standardized volume expansion, a first set of echocardiographic measurements will be performed. Then, we will perform 15-second end-expiratory and end-inspiratory occlusions. Occlusions will be separated by 1 minute to allow the cardiac index to return to its baseline value. A last set of measurements will be performed after fluid administration. Ventilatory settings and other treatments will remain unchanged during the study period.

SUMMARY:
Initial fluid resuscitation remains the first treatment step for most children experiencing circulatory failure and/or systemic hypotension. Only one-half of these patients respond to fluid administration by a significant increase in cardiac output. A positive fluid balance is a poor prognostic factor that increases mortality. There are few markers validated in children to assess volume reactivity by dynamic ultrasound parameters mainly based on heart-lung interaction.

In this work, the investigators propose to investigate whether dynamic parameters validated in adults, such as the superior vena caval collapsibility and the variability of cardiac output during an end-expiratory and end-inspiratory occlusion, are also reliable indicators of volume responsiveness in sedated children under controlled-mode ventilation.

DETAILED DESCRIPTION:
After standardized volume expansion, patients who present an increase of cardiac index measured by transthoracic echocardiography greater than or equal to 15% of baseline measurement will be considered responders .

A previous similar study using respiratory variations in aortic blood flow to predict fluid responsiveness in ventilated children reported a ROC curve area 0.85, while the prevalence rate of circulatory failure was 50%. Given these assumptions, a sample size of 38 subjects per group (Responders / No responders) was estimated to provide a AUC equivalent. A total of 76 subjects should be included.

ELIGIBILITY:
Inclusion Criteria :

* Patient < 18 years (child and neonate)
* Sedated and mechanically ventilated under controlled-mode ventilation
* In whom fluid administration was planned by the attending physicians

Exclusion Criteria :

* High-frequency oscillatory ventilation
* Cardiac arrhythmia
* Congenital heart defect

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 76 (Estimated)
Dates: Start 2021-06-25 (Actual); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Cardiac index measured by transthoracic echocardiography | Through the end of the hospitalisation, a maximum of 2 months
  After fluid administration, patients who present an increase of cardiac index measured by transthoracic echocardiography greater than or equal to 15% of baseline measurement will be considered responders .

SECONDARY OUTCOMES:
End-tidal carbon dioxide levels | Through the end of the hospitalisation, a maximum of 2 months
  ETCO2 measurements using sidestream microstream technology before and after fluid administration will be compared to cardiac index measured by transthoracic echocardiography, ETCO2 increment of 5% is expected in responders patients.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Barreault, Doctor, Principal Investigator — Bicetre Hospital (AP-HP)
Locations (1):
- Bicetre Hospital, Le Kremlin-Bicêtre, France

REFERENCES:
- [Background] Durand P, Chevret L, Essouri S, Haas V, Devictor D. Respiratory variations in aortic blood flow predict fluid responsiveness in ventilated children. Intensive Care Med. 2008 May;34(5):888-94. doi: 10.1007/s00134-008-1021-z. Epub 2008 Feb 8. PMID 18259726